CLINICAL TRIAL: NCT03445442
Title: Different Surgical Techniques Used for Prolapse Repair in Elderly Patient
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: URO-BASE02
Record Dates: First submitted 2018-02-12; First posted 2018-02-26 (Actual); Last update posted 2018-03-22 (Actual); Status verified 2018-02

CONDITIONS: Unrecognized Condition
Keywords: Elderly; Native tissue repair; Pelvic Organ Prolapse; Sacrocolpopexy; Vaginal mesh repair
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1: Sacrocolpopexy (SCP)
  Interventions: Procedure: SCP
- Group 2: Native tissue repair surgery (NTR)
  Interventions: Procedure: NTR
- Group 3: Vaginal mesh repair surgery (VMR)
  Interventions: Procedure: VMR

INTERVENTIONS:
Procedure: SCP — Sacrocolpopexy (SCP) aims to secure the anterior vaginal wall, the uterus more or less the posterior vaginal wall using polypropylene prostheses and to secure them to the presacral ligament to restore the patient's anatomical features and improve pelvic symptoms
  Groups: Group 1
Procedure: NTR — Native tissue repair surgery (NTR) consist of site-specific surgical repair of the existing defect (anterior and/or posterior) using non-absorbable sutures. Specifically, anterior and/or posterior colporrhaphy for cystocele and rectocele respectively after adequate hydrodissection of the vesicovaginal or rectovaginal space.
  Groups: Group 2
Procedure: VMR — Vaginal mesh repair surgery (VMR) is performed using a single-incision mesh system. A single vertical incision is made in the anterior and/or posterior vaginal wall. A full-thickness dissection is performed laterally and apically to the ischial spine.
  Groups: Group 3

SUMMARY:
The investigator aimed to compare various pelvic floor repairs in female aged from 70 to 80 years old, to see which procedure in terms of treatment-related complications of SCP, VMR and NTR by comparing the operative and functional outcomes in this patient population.

DETAILED DESCRIPTION:
Pelvic organ prolapse (POP) is a global health care issue that could have a significant impact on pelvic floor function and quality of life (QOL), while seldom having the potential to be life-threatening. Prevalence of POP increases with age. In women older than 80, 11% undergo a surgical procedure. The incidence of degenerative diseases and multiple co-morbidities increases with age, and advanced age is also associated with an increase in morbidity generally for gynecologic procedures. Furthermore, greater comorbidity beforehand can predispose patients to postoperative complications such as bleeding, hematoma, pain, infectious. As a result hospital stays are longer and the surgical results are compromised.

Surgical techniques should optimize functional results and minimize complications. In POP surgery, younger women are good candidates for sacrocolpopexy (SCP), because of the improved long term functional result, while women older than 80 may have a satisfactory outcome with fewer complication with a vaginal repair with mesh (VMR) or native tissue (NTR). The increasing prevalence of POP, and the increasing population of women aged 70-80 requires an evaluation of the appropriate surgical management since women in this age group may be candidates for all types of surgical repair.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a pelvic organ prolapse
* Patients aged between 70 and 80 years old
* Patients with symptomatic anterior, apical and/or posterior compartment prolapse, stage 2 or greater

Exclusion Criteria:

* Patients with a previous history of pelvic surgery for a cancer diagnosis are excluded
* Patients with a surgical repair specific to the existing defect site (For group 2)

Ages: 70 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The study cohort is selected from our institution. The study involves elderly females over 70 years old with advanced pelvic organ prolapse.
Sampling Method: Non-Probability Sample
Enrollment: 214 (Actual)
Dates: Start 2011-01-01 (Actual); Primary Completion 2012-12-01 (Actual); Study Completion 2017-04-05 (Actual)

PRIMARY OUTCOMES:
Post-operative complications | 12 months follow-up
  All complications are recorded, corresponding to Clavien Dindo classification.

SECONDARY OUTCOMES:
Anatomical success rate | 12 months follow-up
  Assessed by recovery time and anatomical correction
Surgical satisfaction | 12 months follow-up
  Assessed by the validated Surgical Satisfaction Questionnaire (SSQ-8)

IPD SHARING:
Plan to Share IPD: No
CFU, Publication at the European Journal in February 2018

REFERENCES:
- [Background] Samuelsson EC, Victor FT, Tibblin G, Svardsudd KF. Signs of genital prolapse in a Swedish population of women 20 to 59 years of age and possible related factors. Am J Obstet Gynecol. 1999 Feb;180(2 Pt 1):299-305. doi: 10.1016/s0002-9378(99)70203-6. PMID 9988790
- [Background] Gomelsky A, Penson DF, Dmochowski RR. Pelvic organ prolapse (POP) surgery: the evidence for the repairs. BJU Int. 2011 Jun;107(11):1704-19. doi: 10.1111/j.1464-410X.2011.10123.x. PMID 21592280
- [Background] Williams-Russo P, Sharrock NE, Mattis S, Szatrowski TP, Charlson ME. Cognitive effects after epidural vs general anesthesia in older adults. A randomized trial. JAMA. 1995 Jul 5;274(1):44-50. PMID 7791257
- [Background] Luber KM, Boero S, Choe JY. The demographics of pelvic floor disorders: current observations and future projections. Am J Obstet Gynecol. 2001 Jun;184(7):1496-501; discussion 1501-3. doi: 10.1067/mob.2001.114868. PMID 11408873
- [Background] Stepp KJ, Barber MD, Yoo EH, Whiteside JL, Paraiso MF, Walters MD. Incidence of perioperative complications of urogynecologic surgery in elderly women. Am J Obstet Gynecol. 2005 May;192(5):1630-6. doi: 10.1016/j.ajog.2004.11.026. PMID 15902169
- [Background] Tabata T, Yamawaki T, Ida M, Nishimura K, Nose Y, Yabana T. Clinical value of dilatation and curettage for abnormal uterine bleeding. Arch Gynecol Obstet. 2001 Jan;264(4):174-6. doi: 10.1007/s004040000100. PMID 11205702
- [Background] Hornemann A, Kamischke A, Luedders DW, Beyer DA, Diedrich K, Bohlmann MK. Advanced age is a risk factor for higher grade perineal lacerations during delivery in nulliparous women. Arch Gynecol Obstet. 2010 Jan;281(1):59-64. doi: 10.1007/s00404-009-1063-7. Epub 2009 Mar 31. PMID 19333610
- [Background] Sabbagh R, Mandron E, Piussan J, Brychaert PE, Tu le M. Long-term anatomical and functional results of laparoscopic promontofixation for pelvic organ prolapse. BJU Int. 2010 Sep;106(6):861-6. doi: 10.1111/j.1464-410X.2009.09173.x. Epub 2010 Jan 19. PMID 20089111
- [Background] Gerten KA, Markland AD, Lloyd LK, Richter HE. Prolapse and incontinence surgery in older women. J Urol. 2008 Jun;179(6):2111-8. doi: 10.1016/j.juro.2008.01.089. PMID 18423726
- [Background] Visco AG, Wei JT, McClure LA, Handa VL, Nygaard IE; Pelvic Floor Disorders Network. Effects of examination technique modifications on pelvic organ prolapse quantification (POP-Q) results. Int Urogynecol J Pelvic Floor Dysfunct. 2003 Jun;14(2):136-40. doi: 10.1007/s00192-002-1030-3. Epub 2003 Mar 28. PMID 12851759
- [Background] Giuly J, Cravello L, D'Ercole C, Roger V, Porcu G, Blanc B. [Richter's spinofixation in vaginal prolapse]. Chirurgie. 1997;122(7):430-4. French. PMID 9588065
- [Background] Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg. 2004 Aug;240(2):205-13. doi: 10.1097/01.sla.0000133083.54934.ae. PMID 15273542
- [Background] Murphy M, Sternschuss G, Haff R, van Raalte H, Saltz S, Lucente V. Quality of life and surgical satisfaction after vaginal reconstructive vs obliterative surgery for the treatment of advanced pelvic organ prolapse. Am J Obstet Gynecol. 2008 May;198(5):573.e1-7. doi: 10.1016/j.ajog.2007.12.036. PMID 18455537
- [Background] King SW, Jefferis H, Jackson S, Marfin AG, Price N. Laparoscopic uterovaginal prolapse surgery in the elderly: feasibility and outcomes. Gynecol Surg. 2017;14(1):2. doi: 10.1186/s10397-017-1000-x. Epub 2017 Apr 11. PMID 28479877
- [Background] Sung VW, Weitzen S, Sokol ER, Rardin CR, Myers DL. Effect of patient age on increasing morbidity and mortality following urogynecologic surgery. Am J Obstet Gynecol. 2006 May;194(5):1411-7. doi: 10.1016/j.ajog.2006.01.050. PMID 16647926
- [Background] Leung JM, Dzankic S. Relative importance of preoperative health status versus intraoperative factors in predicting postoperative adverse outcomes in geriatric surgical patients. J Am Geriatr Soc. 2001 Aug;49(8):1080-5. doi: 10.1046/j.1532-5415.2001.49212.x. PMID 11555070
- [Background] Maher C, Feiner B, Baessler K, Christmann-Schmid C, Haya N, Brown J. Surgery for women with apical vaginal prolapse. Cochrane Database Syst Rev. 2016 Oct 1;10(10):CD012376. doi: 10.1002/14651858.CD012376. PMID 27696355
- [Background] Rodgers A, Walker N, Schug S, McKee A, Kehlet H, van Zundert A, Sage D, Futter M, Saville G, Clark T, MacMahon S. Reduction of postoperative mortality and morbidity with epidural or spinal anaesthesia: results from overview of randomised trials. BMJ. 2000 Dec 16;321(7275):1493. doi: 10.1136/bmj.321.7275.1493. PMID 11118174
- [Background] Greer JA, Northington GM, Harvie HS, Segal S, Johnson JC, Arya LA. Functional status and postoperative morbidity in older women with prolapse. J Urol. 2013 Sep;190(3):948-52. doi: 10.1016/j.juro.2013.03.004. Epub 2013 Mar 6. PMID 23473899
- [Background] Ganatra AM, Rozet F, Sanchez-Salas R, Barret E, Galiano M, Cathelineau X, Vallancien G. The current status of laparoscopic sacrocolpopexy: a review. Eur Urol. 2009 May;55(5):1089-103. doi: 10.1016/j.eururo.2009.01.048. Epub 2009 Feb 4. PMID 19201521
- [Background] Keys T, Campeau L, Badlani G. Synthetic mesh in the surgical repair of pelvic organ prolapse: current status and future directions. Urology. 2012 Aug;80(2):237-43. doi: 10.1016/j.urology.2012.04.008. Epub 2012 May 23. PMID 22626575
- [Background] Belot F, Collinet P, Debodinance P, Ha Duc E, Lucot JP, Cosson M. [Risk factors for prosthesis exposure in treatment of genital prolapse via the vaginal approach]. Gynecol Obstet Fertil. 2005 Dec;33(12):970-4. doi: 10.1016/j.gyobfe.2005.10.023. French. PMID 16324871
- [Background] Maher CF, Feiner B, DeCuyper EM, Nichlos CJ, Hickey KV, O'Rourke P. Laparoscopic sacral colpopexy versus total vaginal mesh for vaginal vault prolapse: a randomized trial. Am J Obstet Gynecol. 2011 Apr;204(4):360.e1-7. doi: 10.1016/j.ajog.2010.11.016. PMID 21306698
- [Background] Agarwala N, Hasiak N, Shade M. Laparoscopic sacral colpopexy with Gynemesh as graft material--experience and results. J Minim Invasive Gynecol. 2007 Sep-Oct;14(5):577-83. doi: 10.1016/j.jmig.2007.03.005. PMID 17848318
- [Background] Su TH, Lau HH, Huang WC, Hsieh CH, Chang RC, Su CH. Single-incision mesh repair versus traditional native tissue repair for pelvic organ prolapse: results of a cohort study. Int Urogynecol J. 2014 Jul;25(7):901-8. doi: 10.1007/s00192-013-2294-5. Epub 2014 Jan 28. PMID 24469775
- [Background] Nieminen K, Hiltunen R, Takala T, Heiskanen E, Merikari M, Niemi K, Heinonen PK. Outcomes after anterior vaginal wall repair with mesh: a randomized, controlled trial with a 3 year follow-up. Am J Obstet Gynecol. 2010 Sep;203(3):235.e1-8. doi: 10.1016/j.ajog.2010.03.030. Epub 2010 May 21. PMID 20494332
- [Background] Moore RD, Miklos JR. Vaginal repair of cystocele with anterior wall mesh via transobturator route: efficacy and complications with up to 3-year followup. Adv Urol. 2009;2009:743831. doi: 10.1155/2009/743831. Epub 2009 Aug 24. PMID 19710939
- [Background] Lee U, Wolff EM, Kobashi KC. Native tissue repairs in anterior vaginal prolapse surgery: examining definitions of surgical success in the mesh era. Curr Opin Urol. 2012 Jul;22(4):265-70. doi: 10.1097/MOU.0b013e32835459bb. PMID 22617056
- [Derived] Tibi B, Vincens E, Durand M, Bentellis I, Salet-Lizee D, Kane A, Gadonneix P, Severac F, Ahallal Y, Chevallier D, Villet R. Comparison of different surgical techniques for pelvic floor repair in elderly women: a multi-institutional study. Arch Gynecol Obstet. 2019 Apr;299(4):1007-1013. doi: 10.1007/s00404-019-05076-1. Epub 2019 Feb 20. PMID 30788571